CLINICAL TRIAL: NCT03283553
Title: Involving Family to Improve Communication in Breast Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: J1735; IRB00129995 (Other: JHMIRB); SAC170001 (Other Grant/Funding Number: Susan G. Komen Breast Cancer Foundation)
Record Dates: First submitted 2017-08-28; First posted 2017-09-14 (Actual); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Active Breast Cancer Treatment
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Checklist; Patient Access to Records

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent Intervention (Experimental): 1.) A one-page paper-pencil agenda setting checklist completed immediately before a regularly scheduled medical oncology visit to elicit and align patient and companion perspectives regarding issues to discuss with the provider, and to stimulate discussion about the role of the companion in the visit, 2.) facilitated registration for the patient portal (for patient and family member, as desired by the patient), and 3.) education (as relevant) on access to doctor's electronic visit notes.
  Interventions: Other: Checklist, MyChart, OpenNotes
- Usual Care (Placebo Comparator): Care as usual with the medical oncologist.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Checklist, MyChart, OpenNotes — 1) Patient-family agenda-setting checklist, 2) Facilitated proxy registration for MyChart, and 3) Education on access to doctor's electronic visit notes.
  Arms: Multicomponent Intervention
Other: Usual Care — Routine medical oncology care
  Arms: Usual Care

SUMMARY:
This study evaluates a multi-component communication intervention in the outpatient setting to strengthen communication among patients being actively treated for breast cancer and their support network of family members and friends. The intervention comprises: 1.) a patient-family agenda-setting checklist completed immediately before a regularly scheduled oncology visit, 2.) facilitated registration for the patient portal (for patient and family member, as desired by the patient), and 3.) education (as relevant) on access to clinician electronic visit notes. The study team will conduct a two-group randomized trial to examine feasibility of the protocol and to compare quality of communication with oncology providers, understanding of patient's cancer, confidence in managing patient's care and satisfaction with cancer care between patient-companion dyads who are in the intervention group (n=60) and patient-companion dyads who receive usual medical oncology care (n=60).

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among survivors in the US. Most patients with breast cancer receive help from family in making complex decisions about treatment, handling logistically demanding care coordination, and managing symptoms and side effects. Although family members (as defined by each patient) play a vital role in cancer care, they are not formally recognized or assessed in care delivery, and their need for information and support is typically unmet. Lack of attention to family in care delivery is an important gap that too often leaves families without adequate information about patient health and treatments. This may prevent families and patients from engaging in open conversations, cause them unnecessary anxiety, and negatively affect the quality of cancer care and delivery.

Communication is particularly important in cancer care, as the optimal course of action is determined through longitudinal discussion of prognosis, treatments, and patient goals, preferences, and concerns. Strategies to improve communication for serious illnesses such as cancer have been developed, but typically target a specific decision, conversation, or setting, most often the inpatient hospital. There is growing agreement that communication among patients, families, and providers should be initiated early and continue throughout the disease trajectory. However, little is known about how to provide both patients and families with access to timely information about patient health and mechanisms to communicate directly with health care providers, as proposed in this study.

The goal of this study is to test a multicomponent intervention to strengthen communication and longitudinal partnerships among women with breast cancer and their family members. Recent work by the study team has demonstrated the feasibility, acceptability, and benefit of intervention components which will be combined into a single model of care. The study team's preliminary studies indicate that clarifying patient and family expectations regarding the role of family and providing family with timely and comprehensive information about patient health (as desired by the patient) leads to more effective family involvement, more frequent patient-family-provider interactions, more patient-centered communication, and greater preparedness to manage care.

This study will evaluate the feasibility of delivering a multicomponent communication intervention in the outpatient setting comprising: 1.) a patient-family agenda-setting checklist completed immediately before a regularly scheduled medical oncology visit with a participating medical oncologist, 2.) facilitated registration for the patient portal (for patient and family member, as desired by the patient), and 3.) education (as relevant) on access to doctor's electronic visit notes. The study will focus on patients who typically attend medical oncology visits with a family member or trusted friend who are already present and involved in communication. This study will enroll up to 132 patients who are on active treatment for breast cancer, up to 132 family member/friend "companions" and up to 14 medical oncology providers. The study team will compare patients and companions who are in the intervention group (n=60 dyads) with patients and companions who are in the control group and receive usual medical oncology care (n=60 dyads). This study will compare quality of communication with medical oncology providers, understanding of patient's cancer, confidence in managing patient's care, satisfaction with cancer care, and symptoms of anxiety after 3 months, 9 months, and 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Medical oncology patient: Established patient of participating medical oncologist greater than 18 years of age, have a diagnosis of early stage or advanced breast cancer, are receiving active systemic therapy (in the form of IV adjuvant systemic therapy if early stage), are English speaking, able to provide informed consent themselves, and identify a family member who they would like to include in their care.
2. Care partner: Family member (e.g. spouse, adult child, parent, adult sibling or other relative) or unpaid friend who regularly accompanies patient to medical oncology visits.
3. Medical oncology provider: Practicing medical oncology provider at a participating clinic who provides care to patients with breast cancer.

Exclusion Criteria:

1. Medical oncology patients: Younger than 18 years, pregnant, not being treated for breast cancer, do not attend medical oncology visits with family member or unpaid friend or unwilling for their family member or unpaid friend to be contacted.
2. Care partner: Paid non-family member who accompanies patient to visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Wolff, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Kimmel Cancer Center - Medical Oncology, Baltimore, Maryland
  - Johns Hopkins Kimmel Cancer Center at Green Spring Station - Medical Oncology, Lutherville, Maryland

IPD SHARING:
Plan to Share IPD: No
This research involves the collection of data and identifying information from approximately 278 diverse study participants including up to 14 medical oncology clinicians, 132 breast cancer patients, and 132 family member or friend companions. The final dataset will include self-reported demographic and health status measures, information from electronic health records, and information about participant experiences. Even though the final dataset will be stripped of identifying information prior to analysis, the study team believes that there remains a possibility of deductive disclosure of subjects. Upon written request from members of the research community, the following resources will be shared: documentation of the process for accessing the study data and constructing the analytic dataset; the codebook for the master analytic dataset; the analytic plan for each study aim; the algorithms used for measurement of outcome variables; surveys and questionnaires.

REFERENCES:
- [Background] Wolff JL, Roter DL, Barron J, Boyd CM, Leff B, Finucane TE, Gallo JJ, Rabins PV, Roth DL, Gitlin LN. A tool to strengthen the older patient-companion partnership in primary care: results from a pilot study. J Am Geriatr Soc. 2014 Feb;62(2):312-9. doi: 10.1111/jgs.12639. Epub 2014 Jan 13. PMID 24417565
- [Background] Wolff JL, Berger A, Clarke D, Green JA, Stametz R, Yule C, Darer JD. Patients, care partners, and shared access to the patient portal: online practices at an integrated health system. J Am Med Inform Assoc. 2016 Nov;23(6):1150-1158. doi: 10.1093/jamia/ocw025. Epub 2016 Mar 28. PMID 27026614
- [Background] Delbanco T, Walker J, Bell SK, Darer JD, Elmore JG, Farag N, Feldman HJ, Mejilla R, Ngo L, Ralston JD, Ross SE, Trivedi N, Vodicka E, Leveille SG. Inviting patients to read their doctors' notes: a quasi-experimental study and a look ahead. Ann Intern Med. 2012 Oct 2;157(7):461-70. doi: 10.7326/0003-4819-157-7-201210020-00002. PMID 23027317
- [Result] Wolff JL, Aufill J, Echavarria D, Heughan JA, Lee KT, Connolly RM, Fetting JH, Jelovac D, Papathakis K, Riley C, Stearns V, Thorner E, Zafman N, Levy HP, Dy SM, Wolff AC. Sharing in care: engaging care partners in the care and communication of breast cancer patients. Breast Cancer Res Treat. 2019 Aug;177(1):127-136. doi: 10.1007/s10549-019-05306-9. Epub 2019 Jun 4. PMID 31165374
- [Derived] Wolff JL, Aufill J, Echavarria D, Blackford AL, Connolly RM, Fetting JH, Jelovac D, Papathakis K, Riley C, Stearns V, Zafman N, Thorner E, Levy HP, Guo A, Dy SM, Wolff AC. A randomized intervention involving family to improve communication in breast cancer care. NPJ Breast Cancer. 2021 Feb 12;7(1):14. doi: 10.1038/s41523-021-00217-9. PMID 33579966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients of participating clinicians who were in active treatment for early stage or advanced breast cancer were mailed letters describing the study 3 weeks before their next scheduled visit. Patients who did not "opt out" by mail were contacted by research staff to discuss study procedures and administer a screening interview.
Period: Patient Participant Flow
Arm/Group | Multicomponent Intervention | Usual Care
Started | 69 | 63
Patient Baseline Interview | 69 | 62
Patient 3-Month Interview | 67 | 60
Patient 9-Month Interview | 63 | 57
Patient 12-Month Interview | 59 | 50
Completed | 59 | 50
Not Completed | 10 | 13
Not completed — Death | 5 | 10
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 1 | 1
Period: Care Partner Participant Flow
Arm/Group | Multicomponent Intervention | Usual Care
Started (Patients and Care Partners were distinctly contacted for baseline and follow up, so the participation of one was not necessarily contingent on the participation of the other.) | 69 | 63
Care Partner Baseline Interview | 69 | 63
Care Partner 3-Month Interview | 69 | 60
Care Partner 9-Month Interview | 64 | 55
Care Partner 12-Month Interview | 59 | 48
Completed | 59 | 48
Not Completed | 10 | 15
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Discontinued because patient death | 5 | 11

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants include 69 dyads (one patient, one care partner) in the intervention arm and 63 dyads (one patient, one care partner) in the usual care arm, for a total of 132 dyads in the study. Baseline participant data for patient and care partner is reported here distinctly, where possible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Multicomponent Intervention | Usual Care | Total
Number analyzed (Participants) | 69 | 63 | 132
Age, Continuous [Mean (Standard Deviation); unit: years]
  Patient age | 55.1 (13.4) | 52.9 (14.5) | 54.1 (13.9)
  Care Partner age | 54.0 (13.79) | 54.0 (13.5) | 54 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Patient sex: Female | 68 | 63 | 131
  Patient sex: Male | 1 | 0 | 1
  Care Partner sex: Female | 28 | 18 | 46
  Care Partner sex: Male | 41 | 45 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Patient Ethnicity: Hispanic or Latino | 4 | 3 | 7
  Patient Ethnicity: Not Hispanic or Latino | 64 | 60 | 124
  Patient Ethnicity: Unknown or Not Reported | 1 | 0 | 1
  Care Partner Ethnicity: Hispanic or Latino | 2 | 3 | 5
  Care Partner Ethnicity: Not Hispanic or Latino | 65 | 60 | 125
  Care Partner Ethnicity: Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Patient Race: American Indian or Alaska Native | 0 | 0 | 0
  Patient Race: Asian | 1 | 2 | 3
  Patient Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Patient Race: Black or African American | 12 | 14 | 26
  Patient Race: White | 55 | 44 | 99
  Patient Race: More than one race | 1 | 3 | 4
  Patient Race: Unknown or Not Reported | 0 | 0 | 0
  Care Partner Race: American Indian or Alaska Native | 0 | 0 | 0
  Care Partner Race: Asian | 1 | 3 | 4
  Care Partner Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Care Partner Race: Black or African American | 11 | 16 | 27
  Care Partner Race: White | 55 | 40 | 95
  Care Partner Race: More than one race | 0 | 0 | 0
  Care Partner Race: Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 63 | 132
Breast Cancer Disease Stage [Count of Participants; unit: Participants]
  Early Stage Breast Cancer | 35 | 37 | 72
  Metastatic Breast Cancer | 34 | 26 | 60

OUTCOME MEASURES:

1. Primary Outcome: Between-group Differences in Patient Complete Illness Understanding at 9-months
Description: Illness understanding was measured by 4 questions regarding knowledge that is considered to be essential to making informed treatment decisions in serious illness, including: 1.) understanding of illness, 2.) knowledge of disease status, 3.) awareness of disease state, and 4.) expectation of duration of life. We summed responses to each item (coded 1 or 0 to reflect the presence or absence of understanding), yielding a score ranging from 0 to 4. Participants with perfect scores reflecting complete illness understanding (4 of 4 correct responses) were compared to all others.
Time Frame: 9 months
Population: The analysis sample includes the 118 patient-care-partner dyads with complete assessments at 9-months.
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 63 | 55
Participants
  Complete Illness Understanding at 9-Months | 42 | 38
  Not Complete Illness Understanding at 9-Months | 21 | 17
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; Complete illness understanding at 9 months was compared to baseline using logistic regression models estimated with generalized estimating equations (GEE) and an exchangeable correlation specification. Each model included group assignment, time (9 months versus baseline), their interaction, and covariates; Test type: Superiority; p = 0.264, Regression, Logistic — P-value represents interaction for differential changes between time point (9 months compared to baseline) and group assignment; Adjusts for baseline patient education, care partner gender, and patient disease stage

2. Primary Outcome: Between-group Differences in Mean Patient Satisfaction With Cancer Care at 9-months
Description: Outcome was measured with the short-form 10-item version of the Family Satisfaction with Cancer Care (FAMCARE) questionnaire, a validated multi-item instrument that was developed to assess family perspective on cancer care. Respondents are asked to rate 10 items that relate to emotional support, personalization of care, support of decision-making, accessibility, and coordination. Response categories include "very satisfied" (2 points), "satisfied" (1 point), or "not satisfied" (0 points), and the 10-items may be summed to yield a total score (range: 0 to 20) with higher scores reflecting greater satisfaction.
Time Frame: 9 months
Population: The analysis sample includes the 118 patient-care-partner dyads with complete assessments at 9-months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 63 | 55
score on a scale | 16.9 (3.9) | 15.4 (5.4)
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; Satisfaction with cancer care at 9 months was compared to baseline using linear regression models with the difference in the score as the outcome and a term for group assignment as the main independent variable; Test type: Superiority; p = 0.555, Regression, Linear — P-value represents the significance of the term for group assignment; Adjusts for baseline patient education, care partner gender, and patient disease stage

3. Primary Outcome: Between-group Differences in Patient Anxiety at 9-months
Description: Outcome was measured using the Generalized Anxiety Disorder 2-item questionnaire (GAD-2), a well-established 2-item instrument that asks about symptoms of anxiety in a two-week recall period from 0 ("not at all") to 3 ("nearly every day"). Full range is 0-6 with higher scores indicating more anxiety. Symptoms of anxiety refer to a cutpoint of 3+ on the GAD-2.
Time Frame: 9 months
Population: The analysis sample includes the 118 patient-care-partner dyads with complete assessments at 9-months.
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 63 | 55
Participants
  Symptoms of Anxiety at 9-Months | 7 | 8
  No Symptoms of Anxiety at 9-Months | 56 | 47
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; Symptoms of anxiety at 9 months were compared to baseline using logistic regression models estimated with generalized estimating equations (GEE) and an exchangeable correlation specification. Each model included group assignment, time (9 months versus baseline), their interaction, and covariates; Test type: Superiority; p = 0.619, Regression, Logistic — P-value represents interaction for differential changes between time point (9 months vs baseline) and group assignment; Adjusts for baseline patient education, care partner gender, and patient disease stage

4. Primary Outcome: Between-group Differences in Care Partner Complete Illness Understanding at 9-months
Description: as for outcome 1
Time Frame: 9 months
Population: The analysis sample includes the 118 patient-care-partner dyads with complete assessments at 9-months.
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 63 | 55
Participants
  Complete Illness Understanding at 9-Months | 44 | 39
  Not Complete Illness Understanding at 9-Months | 19 | 16
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.532, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Adjusts for baseline patient education, care partner gender, and patient disease stage

5. Primary Outcome: Between-group Differences in Care Partner Satisfaction With Cancer Care at 9-months
Description: Outcome was measured with the short-form 10-item version of the FAMCARE (Family Satisfaction with Cancer Care) questionnaire, a validated multi-item instrument that was developed to assess family perspective on cancer care. Respondents are asked to rate 10 items that relate to emotional support, personalization of care, support of decision-making, accessibility, and coordination. Response categories include "very satisfied" (2 points), "satisfied" (1 point), or "not satisfied" (0 points), and the 10-items may be summed to yield a total score (range: 0 to 20) with higher scores reflecting greater satisfaction.
Time Frame: 9 months
Population: The analysis sample includes the 118 patient-care-partner dyads with complete assessments at 9-months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 63 | 55
score on a scale | 15.7 (4.4) | 15.4 (5.5)
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.108, Regression, Linear — P-value represents the significance of the term for group assignment; Adjusts for baseline patient education, care partner gender, and patient disease stage

6. Primary Outcome: Between-group Differences in Care Partner Anxiety at 9-months
Description: as for outcome 3
Time Frame: 9 months
Population: The analysis sample includes the 118 patient-care-partner dyads with complete assessments at 9-months.
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 63 | 55
Participants
  Symptoms of Anxiety at 9-Months | 8 | 10
  No Symptoms of Anxiety at 9-Months | 55 | 45
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.405, Regression, Logistic — P-value represents interaction for differential changes between time point (9 months vs baseline) and group assignment; Adjusts for baseline patient education, care partner gender, and patient disease stage

7. Secondary Outcome: Between-group Differences in Patient Quality of Communication at 9-months
Description: Outcome was measured using the Quality of Communication (QC) Scale, a validated 10-item instrument to assess quality of communication between the participant and the medical oncology team. The scale for each item is from 0 ('Worst you can imagine') to 10 ('Best you can imagine'). Full range is 0-100 with higher scores indicating higher perceived quality of communication.
Time Frame: 9 months
Population: The analysis sample includes the 118 patient-care-partner dyads with complete assessments at 9-months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 63 | 55
units on a scale | 89.8 (11.6) | 88.0 (18.7)
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; Quality of communication at 9 months was compared to baseline using linear regression models with the difference in the score as the outcome and a term for group assignment as the main independent variable; Test type: Superiority; p = 0.412, Regression, Linear — P-value represents the significance of the term for group assignment; Adjusts for baseline patient education, care partner gender, and patient disease stage

8. Secondary Outcome: Between-group Differences in Care Partner Quality of Communication at 9-months
Description: as for outcome 7
Time Frame: 9 months
Population: The analysis sample includes the 118 patient-care-partner dyads with complete assessments at 9-months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 63 | 55
units on a scale | 90.3 (10.3) | 86.2 (15.9)
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.872, Regression, Linear — P-value represents the significance of the term for group assignment; Adjusts for baseline patient education, care partner gender, and patient disease stage

9. Post Hoc Outcome: Between-group Differences in Care Partner Registration for Shared Access to the Patient Portal at 9-months
Description: Care partner registration for shared access to the patient portal was assessed at baseline and nine-months post-enrollment.
Time Frame: 9 months
Population: The analysis sample includes the 118 patient-care-partner dyads with complete assessments at 9-months.
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 63 | 55
Participants
  Care Partner Registered by 9 Months | 49 | 1
  Care Partner Did Not Register by 9 Months | 14 | 54
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; Test type: Superiority; p < 0.001, Fisher Exact; P-value assess between-group differences in proportion of participants who were registered during the 9-month follow up period

10. Post Hoc Outcome: Between-group Differences in Patient Views of Clinical Visit Notes in the Patient Portal at 9-months
Description: Patient portal use was assessed from date and time-stamped interactions reflecting the frequency, timing, and type of patient portal interactions.Use of the patient portal refers to interactions between enrollment and up to 40-weeks post-enrollment.
Time Frame: 9 months
Population: The analysis sample includes the patients who used a patient portal feature at least once during 9 month follow up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 60 | 50
Participants
  Patient Viewed a Clinical Visit Note by 9-months | 38 | 18
  Patient Did Not View a Clinical Visit Note by 9-months | 22 | 32
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; Test type: Superiority; p = 0.003, Fisher Exact; P-value assess between-group differences in proportion of participants who used a patient portal feature at least once during 9-month follow up

11. Post Hoc Outcome: Between-group Differences in Care Partner Views of Clinical Visit Notes in the Patient Portal at 9-months
Description: Patient portal use was assessed from date and time-stamped interactions reflecting the frequency, timing, and type of patient portal interactions. Use of the patient portal refers to interactions between enrollment and up to 40-weeks post-enrollment.
Time Frame: 9 months
Population: The analysis sample includes the care partners who logged in to the patient portal at least once during 9 month follow up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 49 | 1
Participants
  Care Partner Viewed a Clinical Visit Note by 9-months | 30 | 0
  Care Partner Did Not View a Clinical Visit Note by 9-months | 19 | 1
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; Test type: Superiority; p < 0.001, Fisher Exact; [statistical method as in outcome 10, analysis 1]

12. Post Hoc Outcome: Between-group Differences in Patient Exchange of Direct Messages in the Patient Portal at 9-months
Description: as for outcome 11
Time Frame: 9 months
Population: The analysis sample includes the patients who logged in to the patient portal at least once during 9 month follow up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 60 | 50
Participants
  Patient Exchanged a Direct Message by 9-months | 52 | 38
  Patient Did Not Exchange a Direct Message by 9-months | 8 | 12
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; Test type: Superiority; p = 0.128, Fisher Exact — P-value assess between-group differences in proportion of participants who used a patient portal feature at least once during 9-month follow up

13. Post Hoc Outcome: Between-group Differences in Care Partner Exchange of Direct Messages in the Patient Portal at 9-months
Description: as for outcome 11
Time Frame: 9 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Multicomponent Intervention | Usual Care
Number analyzed (Participants) | 49 | 1
Participants
  Care Partner Exchanged a Direct Message by 9-months | 3 | 0
  Care Partner Did Not Exchange a Direct Message by 9-months | 46 | 1
Statistical Analysis 1: Comparison: Multicomponent Intervention vs Usual Care; Test type: Superiority; p = 0.247, Fisher Exact — [p-value comment as in outcome 12, analysis 1]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Assessed for patients only.
Arm/Group | Multicomponent Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 5/69 | 10/63
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/63
Other Adverse Events (participants affected / at risk) | 0/69 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT03283553/Prot_SAP_000.pdf